CLINICAL TRIAL: NCT05780385
Title: Nasotracheal Intubation Vs. Conventional Airway Management in Critically Ill Patients.
Brief Title: Nasotracheal Intubation in Critically Ill.
Acronym: NaTra-P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NaTra-P
Record Dates: First submitted 2023-03-05; First posted 2023-03-22 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-12

CONDITIONS: Tracheal Intubation Morbidity; Critical Care
Keywords: tracheal intubation; airway management; critical care; nasotracheal intubation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nasotracheal intubation (Experimental)
  Interventions: Device: nasotracheal intubation
- orotracheal intubation (Active Comparator)
  Interventions: Device: orotracheal intubation

INTERVENTIONS:
Device: nasotracheal intubation — patients requiring tracheal intubation receive nasotracheal intubation
  Other Names: NTI
  Arms: nasotracheal intubation
Device: orotracheal intubation — patients requiring tracheal intubation receive orotracheal intubation
  Other Names: OTI
  Arms: orotracheal intubation

SUMMARY:
The aim of this prospective randomized trail is to compare nasotracheal versus orotracheal intubation in critically ill patients. We aim to study:

* required sedation depth
* rate of spontaneous breathing
* extend and possibility of physiotherapy
* vasopressor and sedative drug doses

Participants are randomized 1:1 to receive either nasotracheal or orotracheal intubation.

DETAILED DESCRIPTION:
In the intensive care unit endotracheal intubation and consecutive mechanical ventilation are required for different surgical procedures, examinations and interventions in the ICU or due to respiratory insufficiency. Commonly, intubation is performed orotracheally by direct laryngoscopy after preoxygenation and administration of narcotics and a muscle relaxant. When using this technique sedation is often necessary for tolerance of the orotracheal tube. To avoid the adverse side effects of sedation and mechanical ventilation as for example hypotension, barotrauma, ventilator associated pneumonia, etc., intubation via a nasotracheal approach might be favorable. Retrospective data show that nasotracheal intubation is associated with fewer sedatives, vasopressors, and a higher rate of spontaneous breathing. As there is a paucity of data concerning the use of nasotracheal intubation in the intensive care setting the investigators aim to compare the use of orotracheal and nasotracheal tubes in a prospective randomized trial, using sedation depth as primary outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients requiring tracheal intubation during their intensive care stay.

Exclusion Criteria:

* orotracheal or nasotracheal route of intubation technically not possible (e.g. confirmed indication for awake fiberoptic intubation due to expected difficult airway)
* tracheal intubation indicated for deep sedation (e.g. treatment of elevated intracranial pressure)
* thrombocytopenia < 50/nl or other risk factors for bleeding
* pregnant or breastfeeding women
* denial of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Sedation depth | intubation to 72 hours
  fraction of time with a Richmond Agitation and Sedation Scale (RASS) of 0 or -1. Range -5 to +4 with 0 as optimum value representing awake and alert patient.

SECONDARY OUTCOMES:
Sedation depth | intubation to day 10
  fraction of time with Richmond Agitation and Sedation Scale (RASS) above and below targeted RASS of 0 or -1. Range -5 to +4 with 0 as optimum value representing awake and alert patient.
time to extubation | intubation to day 30
  time until airway device can be removed or patient receives tracheostomy
rate of extubation | intubation to day 30
  rate of successful removal of airway device without tracheostomy
tracheostomy | intubation to day 30
  rate of tracheostomy
spontaneous breathing | intubation to day 10
  rate of spontaneous breathing while on airway device
vasopressor therapy | intubation to day 10
  doses of vasopressor drugs while on airway device
sedative drugs | intubation to day 10
  doses of sedative drugs therapy while on airway device
ventilator associated pneumonia | intubation to day 30
  incidence of ventilator associated pneumonia associated with airway device
sinusitis | intubation to day 30
  incidence of sinusitis associated with airway device
physiotherapy | intubation to day 10
  intensive care unit mobility score (ICU-MS), Range 0 to 10 with higher values indicating higher extend of physiotherapy
length of intensive care stay | intubation to day 30
  length of intensive care stay
complications | intubation to day 1
  complications associated with intubation (i.e. bleeding, damage to teeth, aspiration)
mortality | intubation to day 30
  mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jörn Grensemann, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamburg, Germany